CLINICAL TRIAL: NCT02008812
Title: Ad Sensor-based Real-time Diagnosis of Adenovirus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 201108029RD
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Adenovirus
Keywords: Adenovirus
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (1):
- Ad sensor (Experimental): virus detection
  Interventions: Device: Ad sensor

INTERVENTIONS:
Device: Ad sensor — Ad sensor, which was developed for the rapid and sensitive detection of viral antigen in medical samples, will be used for analyzing the interaction kinetics between anti-Adenovirus and its Adenovirus antigen present in patients and normal samples.
  The system incorporates the use of chip formats. In antibody probing, antibodies are bound as a suitable probe, which specifically and selectively binds targeted molecules (virus antigen) in the test specimens.

SUMMARY:
To develop a real-time diagnostic technique with Ad sensor for Adenovirus detection, the investigators conduct a prospective clinical study. In comparison with results from direct sequencing of Adenovirus, the investigators evaluate the performance of Ad sensor , including reproducibility, sensitivity, specificity, and cross-reaction. The potential factors which may interfere with the results would be investigated. With such technique, the investigators hope to make early diagnosis and give Adenovirus patients early treatment to reduce the complications and case-fatality rate.

DETAILED DESCRIPTION:
1. Sample acquirement： At National Taiwan University Hospital in Taiwan, we will enroll patients who have Adenovirus infection . We will take three throat swabs for each patient: one for viral isolation, one for RT-PCR and the last for the Ad sensor - based real-time diagnosis.
2. Ad sensor diagnosis： Ad sensor (structural chip-based optosensing virus probing system), which is for the rapid and sensitive detection of viral antigen in medical samples, will be used for analyzing the interaction kinetics between anti-Adenovirus and its Adenovirus antigen present in patients'and normal samples.
3. Gold standard： viral isolation and RT-PCR

ELIGIBILITY:
Inclusion Criteria:

A: The patients with confirmed or suspected infection. B: The healthy person without disease.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The performance of Ad sensor | 1 Day
  In comparison with results from viral isolation and RT-PCR of Adenovirus , we evaluate the performance of Ad sensor, including sensitivity, specificity, cross-reaction and reproducibility.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan